CLINICAL TRIAL: NCT04425564
Title: Clinico-pharmacological Study of Metronomic Capecitabine and Oxaliplatin Versus Classic XELOX in Egyptian Metastatic Colorectal Cancer
Brief Title: Study of Metronomic Capecitabine and Oxaliplatin Versus XELOX in Egyptian Metastatic Colorectal Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201516007.3
Record Dates: First submitted 2020-06-02; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Clinical Response; Toxicity; Survival
Keywords: colorectal cancer; metronomic capecitabine
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Oxaliplatin; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Classic (A) (Active Comparator): patients recieving classic XELOX (oxaliplatin 130mg/m2 and capecitabine 1000mg/m2 bid)
  Interventions: Drug: Classic XELOX; Other: Blood samples for pharmacological studies
- metronomic (B) (Experimental): patients recieving low dose capecitabine (2000mg daily divided in two doses for 8 weeks) and oxaliplatin (30mg/m2 weekly for eight weeks) followed by 2 weeks rest.
  Interventions: Drug: metronomic XELOX; Other: Blood samples for pharmacological studies

INTERVENTIONS:
Drug: metronomic XELOX
  Other Names: Capecitabine; Oxaliplatin
  Arms: metronomic (B)
Drug: Classic XELOX
  Other Names: Capecitabine; Oxaliplatin
  Arms: Classic (A)
Other: Blood samples for pharmacological studies
  Other Names: No other names

SUMMARY:
Colorectal cancer (CRC) in Egypt is advanced tumors at diagnosis. Although, the dramatic increase in efficacy, reduction of mortality, and improvements in survival by the use of standard doses of chemotherapy, some CRC patients suffer from severe toxicities besides disease progression. Use of chemotherapy less than the maximum tolerated dose, with no prolonged drug free breaks incapacitates the cells to engage in progression mechanisms, suggesting that it could be a better alternative to standard dose therapy with better toxicity profile

DETAILED DESCRIPTION:
This is a randomized phase II prospective study that included 70 (35 in each arm) metastatic Egyptian CRC cancer patients diagnosed at the National Cancer Institute, Cairo University between January 2016 and June 2018). Patients were randomly treated with either classic XELOX (arm A) or with capecitabine (2000 mg daily x 8 weeks) and oxaliplatin (30 mg/m2 weekly X 8 weeks) then 2 weeks rest (arm B). Toxicities and the survival analysis after two years for both regimens were recorded. Blood samples are taken from both groups to assess pharmacokinetics of capecitabine and its relation to dosing.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18-70 years of both sexes.
* PS 0-2 and histologically proven mCRC with unresectable metastases (rectal cancer is included to left side cancers).
* They should have measurable lesions (that can be accurately measured in at least one dimension using calipers or ruler and measurement must be at least 20 mm using conventional techniques or 10 mm using spiral CT scan).
* No previous treatment for metastatic disease and had ended adjuvant treatment > 6 months.
* peripheral neuritis less than grade 2.
* Normal organ functions:(Creatinine ≤1.2, Bilirubin ≤1.2, SGOT/SGPT< 2N, HB >9gm/dl, WBC>3.5/dl with ANC >1.5/dl, Plat ≥100/dl).
* For patients with liver metastases, Bilirubin should not be >2.5N and transaminases not >5N. (All patients were screened for HCV and HBS Ag by PCR).
* Adequate cardiac functions (EF>55%)

Exclusion Criteria:

* patients with only ascites or bone metastasis

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
response rates | two years
  Calculated with 95% confidence interval
Rate of toxicities and grades | two years
  Categorical data summarized by pecentages
Peak and trough levels of capecitabine and relation to dosing | Two years
  Numerical data summarized by means and standard deviation

SECONDARY OUTCOMES:
Progression free survival | two years
  Cox proportional hazard model
Overall survival | Two years
  Kaplan and Meier test

IPD SHARING:
Plan to Share IPD: No